CLINICAL TRIAL: NCT02036242
Title: Sole Epidural Local Anesthetic Versus Opioid Plus Local Anesthetic in Epidural Labor Pain Control
Brief Title: Sole Local Anesthetic Versus Opioid Plus Local Anesthesia in Epidural Labor Analgesia
Acronym: OLAA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Fu Zhou Wang, Dr, Nanjing Medical University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: NJFY13007; JQX12009 (Other Grant/Funding Number: Nanjing Municipal Bureau of Health)
Record Dates: First submitted 2014-01-11; First posted 2014-01-14 (Estimated); Last update posted 2014-02-04 (Estimated); Status verified 2014-02

CONDITIONS: Pain
Keywords: Opioid; Local anesthetic; Labor delivery; Safety
MeSH Terms: conditions — Pain | interventions — Ropivacaine; Sufentanil; Analgesics, Opioid; Anesthetics, Local

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sole local anesthetic (Experimental): Epidural analgesia will be given with sole local anesthetic (0.125% ropivacaine) intermittently
  Interventions: Drug: Sole local anesthetic; Drug: Ropivacaine
- Opioid plus local anesthetic (Active Comparator): Epidural analgesia will be given with opioid (sufentanil) combined with local anesthetic (0.125% ropivacaine) intermittently
  Interventions: Drug: Sufentanil (Opioid plus local anesthetic); Drug: Ropivacaine

INTERVENTIONS:
Drug: Sole local anesthetic — 0.125% ropivacaine 10-15 ml every 1h during labor delivery
  Other Names: Ropivacaine; Naropin
  Arms: Sole local anesthetic
Drug: Sufentanil (Opioid plus local anesthetic) — Sufentanil combined with 0.125% ropivacaine, 10-15 ml every 1h during labor delivery
  Other Names: Naropin
  Arms: Opioid plus local anesthetic
Drug: Ropivacaine

SUMMARY:
It is common for obstetric anesthesia using opioid supplement to local anesthetics for epidural labor pain control. Given the low doses of these epidural drugs, we never doubt the necessity of the supplement of opioid to lacal anesthetics during this process based on the concept that opioid addition can enhance and prolong the analgesic effect of local anesthetics. However, we unavoidably encounter many opioid-associated side effects during the labor delivery. In addition, usage of opioid increase the medical cost for each patient. We herein hypothesized that in the context of obstetric anesthesia, sole local anesthetics can produce as the same analgsic effect as opioid plus local anesthetics given for epidural labor pain control.

ELIGIBILITY:
Inclusion Criteria:

* Nulliparas
* Request epidural analgesia
* Chinese

Exclusion Criteria:

* Allergic to opioid or local anesthetics
* Fail to perform epidural puncture and catheterization
* Organ dysfunction
* Contraindications for epidural anesthesia

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 500 (Actual)
Dates: Start 2013-09; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Pain scorings | up to 3 days
  Using visual analog scale (VAS) assess the pain intensity at the following time points: (1) immediate after randomization; (2) prior to epidural analgesia; (3) 0, 5, 10, 30, 60 min after epidural analgesia; (4) every 1 h for VAS pain 60 min later after epidural analgesia; (5) at cervical dilation reach to 4 cm and 10 cm; (6) when pushing starts; (7) after completion of labor; (8) post-delivery days 1, 2 and 3.

SECONDARY OUTCOMES:
Pruritus | From post-randomization to post-delivery day 3
  Record incidence of pruritus at the following time points: (1) immediate after randomization; (2) prior to epidural analgesia; (3) 0, 5, 10, 30, 60 min after epidural analgesia; (4) every 1 h 60 min later after epidural analgesia; (5) at cervical dilation reach to 4 cm and 10 cm; (6) when pushing starts; (7) after completion of labor; (8) post-delivery days 1, 2 and 3.
Dizziness | From post-randomization to post-delivery day 3
  Record incidence of dizziness at the following time points: (1) immediate after randomization; (2) prior to epidural analgesia; (3) 0, 5, 10, 30, 60 min after epidural analgesia; (4) every 1 h 60 min later after epidural analgesia; (5) at cervical dilation reach to 4 cm and 10 cm; (6) when pushing starts; (7) after completion of labor; (8) post-delivery days 1, 2 and 3.
Nausea | From post-randomization to post-delivery day 3
  Record incidence of nausea at the following time points: (1) immediate after randomization; (2) prior to epidural analgesia; (3) 0, 5, 10, 30, 60 min after epidural analgesia; (4) every 1 h 60 min later after epidural analgesia; (5) at cervical dilation reach to 4 cm and 10 cm; (6) when pushing starts; (7) after completion of labor; (8) post-delivery days 1, 2 and 3.
Vomiting | From post-randomization to post-delivery day 3
  Record incidence of vomiting at the following time points: (1) immediate after randomization; (2) prior to epidural analgesia; (3) 0, 5, 10, 30, 60 min after epidural analgesia; (4) every 1 h 60 min later after epidural analgesia; (5) at cervical dilation reach to 4 cm and 10 cm; (6) when pushing starts; (7) after completion of labor; (8) post-delivery days 1, 2 and 3.
Drowsiness | From post-randomization to post-delivery day 3
  Record incidence of drowsiness at the following time points: (1) immediate after randomization; (2) prior to epidural analgesia; (3) 0, 5, 10, 30, 60 min after epidural analgesia; (4) every 1 h 60 min later after epidural analgesia; (5) at cervical dilation reach to 4 cm and 10 cm; (6) when pushing starts; (7) after completion of labor; (8) post-delivery days 1, 2 and 3.
Sedation | From post-randomization to post-delivery day 3
  Record incidence of sedation at the following time points: (1) immediate after randomization; (2) prior to epidural analgesia; (3) 0, 5, 10, 30, 60 min after epidural analgesia; (4) every 1 h 60 min later after epidural analgesia; (5) at cervical dilation reach to 4 cm and 10 cm; (6) when pushing starts; (7) after completion of labor; (8) post-delivery days 1, 2 and 3.
Respiratory depression | From post-randomization to post-delivery day 3
  Record incidence of respiratory depression at the following time points: (1) immediate after randomization; (2) prior to epidural analgesia; (3) 0, 5, 10, 30, 60 min after epidural analgesia; (4) every 1 h 60 min later after epidural analgesia; (5) at cervical dilation reach to 4 cm and 10 cm; (6) when pushing starts; (7) after completion of labor; (8) post-delivery days 1, 2 and 3.
Psychological effects | From post-randomization to post-delivery day 3
  Record incidence of psychological effects [euphoria, hallucinations, delirium and confusion] at the following time points: (1) immediate after randomization; (2) prior to epidural analgesia; (3) 0, 5, 10, 30, 60 min after epidural analgesia; (4) every 1 h 60 min later after epidural analgesia; (5) at cervical dilation reach to 4 cm and 10 cm; (6) when pushing starts; (7) after completion of labor; (8) post-delivery days 1, 2 and 3.
Myoclonus | From post-randomization to post-delivery day 3
  This describes muscle rigidity and abnormal movement of the limbs and muscles.
  Record incidence of myoclonus at the following time points: (1) immediate after randomization; (2) prior to epidural analgesia; (3) 0, 5, 10, 30, 60 min after epidural analgesia; (4) every 1 h 60 min later after epidural analgesia; (5) at cervical dilation reach to 4 cm and 10 cm; (6) when pushing starts; (7) after completion of labor; (8) post-delivery days 1, 2 and 3.
Maternal heart rate | From post-randomization to post-delivery day 3
  Record incidence of maternal heart rate at the following time points: (1) immediate after randomization; (2) prior to epidural analgesia; (3) 0, 5, 10, 30, 60 min after epidural analgesia; (4) every 1 h 60 min later after epidural analgesia; (5) at cervical dilation reach to 4 cm and 10 cm; (6) when pushing starts; (7) after completion of labor; (8) post-delivery days 1, 2 and 3.
Miosis | From post-randomization to post-delivery day 3
  Record incidence of miosis at the following time points: (1) immediate after randomization; (2) prior to epidural analgesia; (3) 0, 5, 10, 30, 60 min after epidural analgesia; (4) every 1 h 60 min later after epidural analgesia; (5) at cervical dilation reach to 4 cm and 10 cm; (6) when pushing starts; (7) after completion of labor; (8) post-delivery days 1, 2 and 3.
Cesarean section | The time at the end of the labor delivery
  Record the incidence of Cesarean section after completion of the labor delivery.

OTHER OUTCOMES:
Time to latent phase | From the beginning of regular contraction of uterus to the dilation of cervical 4cm
  Record the time duration
Time of active phase | From the cervix 4cm to the dilation of cervical 10cm
  Record the time duration
Overall satisfaction of analgesia | At the time of the end of the labor delivery
  Assess the analgesia satisfaction after the completion of the labor delivery
Oxytocin usage | At the time of the end of the labor
  Record the total usage of oxytocin after completion of the labor delivery
Neonatal Apgar score | At the time of the baby was born, 1min, 5min, 10min and 20min
Instrumental delivery | At the time of the end of the labor
  Record the incidence of instrumental delivery after completion of the labor delivery.
Umbilical gas analysis | At the time of the fetus was delivery

CONTACTS AND LOCATIONS:
Locations (1):
- Nanjing Maternity and Child Health Care Hospital, Nanjing, Jiangsu, China

REFERENCES:
- [Derived] Wang X, Xu S, Qin X, Li X, Feng SW, Liu Y, Wang W, Guo X, Shen R, Shen X, Wang F. Comparison Between the Use of Ropivacaine Alone and Ropivacaine With Sufentanil in Epidural Labor Analgesia. Medicine (Baltimore). 2015 Oct;94(43):e1882. doi: 10.1097/MD.0000000000001882. PMID 26512604